CLINICAL TRIAL: NCT07301099
Title: Epidemiology and Current Practices in Severe Community-Acquired Pneumonia (PLENITUDE)
Brief Title: Epidemiology and Current Practices in Severe Community-Acquired Pneumonia
Acronym: PLENITUDE
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad de la Sabana (Other)
Collaborators: International Severe Acute Respiratory and Emerging Infection Consortium (Other); European Society of Intensive Care Medicine (Other); Latin American Intensive Care Network (LIVEN) (Unknown)
Responsible Party: Sponsor
Other Study IDs: Acta No. 690 10-Oct-2025; 20251004 (Other: Clínica Universidad de La Sabana)
Record Dates: First submitted 2025-12-15; First posted 2025-12-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Severe Community-acquired Pneumonia (sCAP)
Keywords: Pneumonia; Respiratory Tract Infections; Community-Acquired Pneumonia; Respiratory Tract Diseases
MeSH Terms: conditions — Community-Acquired Pneumonia; Pneumonia; Respiratory Tract Infections; Respiratory Tract Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Lower respiratory tract sample (either sputum or endotracheal aspirates) for conventional culture, multiplex PCR testing (virus and/or bacterial detection)
  * Blood and urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients with Severe Community-Acquired Pneumonia (sCAP): Clinical follow-up for 12 months

SUMMARY:
The goal of this observational study is to learn more about severe community-acquired pneumonia (sCAP) in adults who need hospital or intensive care. This type of pneumonia starts outside the hospital and can quickly become life-threatening. The study aims to understand how people with sCAP are cared for in different parts of the world and how these differences relate to their recovery.

* The main questions this study aims to answer are:
* What are the characteristics, treatments, and outcomes of adults with sCAP?
* How closely do hospitals follow international guidelines for diagnosing and treating sCAP?
* What factors are linked to worse outcomes, such as the need for a ventilator or risk of death?

This study will not test any new drugs or procedures. Instead, researchers will observe the care that participants already receive as part of their normal treatment. Hospitals in many countries will take part, including centres in Europe, North America, Latin America, Asia, Africa, and Oceania. This global participation will help show how sCAP affects people in different health systems and communities.

Participants will be adults who arrive at a hospital or intensive care unit with severe pneumonia. Most information will come from medical records, such as symptoms, test results, treatments given, and how participants respond to care. In some hospitals with special laboratory capacity, additional blood or breathing samples may be collected to study how the body fights infection.

No extra visits are required for routine data-only participants. In sites that collect samples, these will usually be taken at the same time as routine medical care to avoid extra procedures. Researchers will also ask about recovery after hospital discharge at 60 days, 6 months, and 12 months. These follow-ups will help us understand long-term health, complications, and quality of life after sCAP.

By collecting information from a large number of hospitals around the world, this study hopes to identify patterns that can help improve diagnosis, treatment, and survival for people with severe pneumonia. The findings may also help health care teams and public health leaders update treatment guidelines and strengthen care for future patients.

DETAILED DESCRIPTION:
Severe community-acquired pneumonia (sCAP) is a life-threatening infection requiring hospital or ICU care. Mortality remains high, and there are major differences worldwide in diagnosis, treatment practices, and availability of resources. Although new international guidelines exist, real-world implementation is not well understood. The PLENITUDE study is a multinational, prospective observational cohort designed to describe global practices, outcomes, microbiology, and biological responses in adults with sCAP using a harmonized research framework.

The study uses a tiered approach aligned with the ISARIC/WHO Clinical Characterisation Protocol. Tier 0 sites collect standardized clinical data from routine medical records. Tier 1 sites also collect a single set of biological samples at admission. Tier 2 sites perform serial biological sampling to evaluate pathogen dynamics and host immune responses over time. This structure allows participation from hospitals with varying levels of resources while preserving core standardization.

Data are collected using variables derived from the ISARIC ARC library to ensure consistency across regions. Clinical information includes demographics, comorbidities, illness severity, laboratory and imaging results, respiratory support, microbiology, treatments, complications, and outcomes. All data are entered into a secure REDCap platform with automated validation rules, range checks, and logic checks. Participant confidentiality is maintained through unique study identifiers and restricted access for authorized personnel.

Quality assurance procedures include programmed data validation, periodic monitoring of completeness and protocol adherence, and selective source data verification. Standard Operating Procedures guide patient identification, sample handling, data entry, and reporting of deviations. Site teams receive training in protocol operations and data management.

Tier 1 and Tier 2 samples follow standardized processing steps based on the ISARIC/WHO CCP, including centrifugation, aliquoting, freezing, and safe handling according to biosafety requirements. Regional laboratory hubs support advanced analyses such as molecular pathogen detection, sequencing, and immune response profiling, improving comparability and quality control across participating countries.

The statistical analysis plan includes descriptive summaries of clinical presentation and management, comparative analyses across regions or guideline adherence groups, multivariable models for risk factor identification, time-to-event analyses, and mixed-effects models for repeated measures in Tier 2. Unsupervised clustering will be used to explore phenotypes and endotypes. Missing data will be addressed using multiple imputation and sensitivity analyses.

Participants are followed during hospitalization and after discharge at 60 days, 6 months, and 12 months to evaluate long-term outcomes, readmissions, persistent symptoms, and quality of life. Follow-up methods include record review and phone or electronic assessments, depending on site capability.

The study is overseen by international Principal Investigators, a Steering Committee of experts, and a centralized data management team. PLENITUDE is expected to generate real-world evidence on global sCAP management, guideline adherence, microbial and immune patterns, and long-term outcomes. These findings may inform improvements in clinical care, strengthen public health strategies, and support future advances in precision medicine for severe pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older are hospitalised with a clinical diagnosis of sCAP according to the American Thoracic Society/Infectious Diseases Society of America (ATS/IDSA) criteria.16
* Admission to participating hospitals or ICUs during the study period.
* Provision of informed consent by the patient or legally authorised representative for those centres collecting biological samples. Data-only participants will not be required to sign informed consent.

Exclusion Criteria:

* Paediatric population (<18 years old)
* Pneumonia acquired in the hospital setting (i.e., nosocomial or hospital-acquired pneumonia).
* Insufficient clinical information to confirm the diagnosis of sCAP.
* Immunosuppression: i.e. Active cancer, hematopoietic cell transplant, solid organ transplant recipients, HIV diagnosed patients regardless of CD4 cell count, chronic immunosuppression with corticosteroids, inborn errors of immunity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enrol adult patients presenting with severe community-acquired pneumonia (sCAP) at participating hospitals and intensive care units worldwide. Participants will be identified through routine clinical care upon hospital or ICU admission. The study includes centres across Europe, North America, Latin America, Asia, Africa, and Oceania, ensuring broad geographical and healthcare system representation. Data-only participants will be sourced from electronic medical records, while biological samples will be collected in Tier 1 and Tier 2 sites with laboratory capacity. The multinational design allows inclusion of patients from high-, middle-, and low-income countries, supporting a diverse and globally representative cohort.
Sampling Method: Non-Probability Sample
Enrollment: 2588 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
All-Cause In-Hospital Mortality | From hospital admission to hospital discharge (up to 30 days)
  Proportion of enrolled adult patients with severe community-acquired pneumonia (sCAP) who die from any cause during the index hospitalisation. Mortality status will be abstracted from clinical and administrative records at ICU and hospital discharge. This measure describes the severity and outcomes of sCAP across diverse international healthcare settings.
Adherence to International sCAP Management Guidelines | During the index hospitalisation (up to 30 days)
  Percentage of adherence to the ERS/ESICM/ESCMID/ALAT guidelines for the management of severe community-acquired pneumonia. Adherence will be quantified using predefined key indicators related to diagnostic evaluation, antibiotic initiation, ventilatory support, biomarker use, ICU management and follow-up practices. This measure evaluates real-world implementation of guideline-based care across participating centres.

SECONDARY OUTCOMES:
ICU Mortality | From ICU admission to ICU discharge (up to 30 days)
  Proportion of patients with sCAP who die during the ICU stay. Mortality status will be obtained from clinical and administrative records. This outcome allows comparison of mortality patterns across regions and centres and contributes to understanding the severity and progression of sCAP within critical care settings.
60-Day and 180-Day Mortality | 60 days and 180 days after enrolment
  Proportion of enrolled patients who die within 60 and 180 days after hospital admission. Mortality will be assessed through clinical records, follow-up contacts, and post-discharge documentation. This outcome characterises mid- and long-term survival trajectories in patients who experience sCAP.
Length of Hospital Stay | From hospital admission to discharge (up to 30 days)
  Number of days from hospital admission to discharge or death. This measure reflects clinical severity, resource utilisation, and recovery trajectory across diverse healthcare settings.
Duration of Mechanical Ventilation | During the index hospitalisation (up to 30 days)
  Total duration (in days) of invasive or non-invasive mechanical ventilation among patients requiring respiratory support. This outcome provides insight into respiratory failure severity and treatment practices across participating ICUs.
Occurrence of Major Complications | During the index hospitalisation (up to 30 days)
  Proportion of patients experiencing complications such as septic shock, ARDS, secondary infections, or multi-organ failure during hospitalisation. Complications will be identified using predefined clinical criteria abstracted from medical records.
ICU or Hospital Readmission | 60 days and 180 days after discharge
  Proportion of patients readmitted to the ICU or hospital within 60 or 180 days after discharge. Readmissions will be assessed through clinical documentation, follow-up visits, and contact with participants or family members.
Health-Related Quality of Life (HRQoL) | At hospital discharge (assessed up to 90 days from admission), and at 12 months (±30 days) following hospital discharge.
  Assessment of Health-Related Quality of Life (HRQoL) using the validated EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) at the day of hospital discharge and during follow-up evaluation at 12 months post-discharge. This outcome aims to quantify long-term functional recovery and wellbeing after severe community-acquired pneumonia (sCAP).

CONTACTS AND LOCATIONS:
Overall Officials: Luis Felipe Reyes, MD, MSc, PhD, Principal Investigator — Universidad de la Sabana; Ignacio-Martin Loeches, MD, PhD, FJFICMI, Principal Investigator — St James's Hospital, Trinity College Dublin
Locations (1):
- Clínica Universidad de La Sabana, Chía, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding the sharing of individual participant data has not yet been finalized. IPD availability will depend on ethical approvals, institutional policies, and data-governance requirements across participating sites.